CLINICAL TRIAL: NCT06782425
Title: A Single-center, Single-arm, Dose-escalation Exploratory Clinical Trial of the Safety, Efficacy, and Pharmacokinetics of XKDCT225 (Targeting Claudin18.2-CAR-T) Cell Injectionin Claudin18.2-positive Advanced Solid Tumors
Brief Title: Treating Claudin18.2-positive Advanced Solid Tumors with XKDCT225(Targeting Claudin18.2-CAR-T)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen Celconta Life Science Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023YP30H02
Record Dates: First submitted 2025-01-02; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Claudin18.2 Positive Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Autologous targeted claudin18.2 chimeric antigen receptor T cell injection (Experimental): Autologous targeted claudin18.2 chimeric antigen receptor T cell injection
  Interventions: Drug: XKDCT225

INTERVENTIONS:
Drug: XKDCT225 — Autologous targeted claudin18.2 chimeric antigen receptor T cell injection

SUMMARY:
A single-center, single-arm, dose-escalation exploratory clinical trial of the safety, efficacy, and pharmacokinetics of XKDCT225 cell injection in Claudin18.2-positive advanced solid tumors

DETAILED DESCRIPTION:
This study is a prospective, single-arm, open-label, single-dose dose-finding study to evaluate the safety, tolerability, pharmacokinetics, and anti-tumor efficacy characteristics of XKDCT225 cell injection preparation in subjects with Claudin18.2-positive advanced solid tumors.

The study will enroll subjects with pathologically confirmed advanced solid tumors, positive Claudin18.2 expression, who have previously received standard treatment, failed treatment or cannot tolerate it. Imaging examinations show evaluable tumor lesions.

This study adopts a single-arm, single-center, dose-escalation design, and uses "accelerated titration" and "3+3" trial designs for dose escalation . It is expected to include 9-18 patients to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of XKDCT225 cell injection .

Main purpose:

the safety and tolerability of XKDCT225 cell injection in patients with Claudin18.2-positive advanced solid malignancies.

Secondary Purpose:

the pharmacokinetic and pharmacodynamic characteristics of XKDCT225 cell injection in patients with Claudin18.2-positive advanced solid malignancies; To preliminarily evaluate the efficacy of XKDCT225 cell injection in patients with Claudin18.2-positive advanced solid malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 (including the critical value), regardless of gender;
2. Patients with advanced solid tumors (including but not limited to gastric adenocarcinoma, esophagogastric junction adenocarcinoma, esophageal adenocarcinoma) with moderate to high expression of Claudin18.2 (expression intensity ≥ 2+ and tumor cell positive rate ≥ 50 %), and whose condition cannot be completely relieved or continues to progress after adequate treatment;
3. At least one measurable lesion according to RECIST 1.1 criteria (non-lymph node lesion with long diameter ≥10 mm, lymph node lesion with short diameter ≥15 mm);
4. Estimated life expectancy > 12 weeks;
5. ECOG physical status score 0 ~ 1;
6. Laboratory test values for screening must meet the following criteria:

Routine blood test:

* WBC≥3.0×10^9 /L
* ANC≥1.5×10^9 /L
* LYMPH≥0.5×10^9 /L
* HB≥90g/L
* PLT≥75×10^9 /L

Blood biochemistry examination:

* ALT and AST ≤ 2.5 × ULN (≤ 5 × ULN if liver metastasis is present)
* ALB≥30g/L
* Serum creatinine ≤1.5×ULN or GFR>50mL/min (GFR = [(140-age)×weight×(0.85female)]/(72×Scr))
* TBIL≤1.5×ULN

Coagulation function test:

* APTT ≤ 1.5 ULN, with INR or PT ≤ 1.5 ULN (not receiving anticoagulation therapy) 7. Female subjects of childbearing age must undergo a serum pregnancy study with negative results at screening and before purging, and be willing to use medically approved highly effective contraceptive methods during the study and for at least 1 year after the last study treatment. Male subjects whose partners are female subjects of childbearing age should undergo surgical sterilization or agree to use effective contraceptive methods during the study and for at least 1 year after the last study treatment, and are prohibited from donating sperm within 1 year.

  8. If the patient is using the following medications, the corresponding conditions must be met:
* Steroids: Therapeutic doses of steroids must be discontinued 4 weeks prior to XKDCT 225 cell injection. However, physiological replacement doses of steroids are allowed: hydrocortisone or equivalent <6~ 12mg / mm^2 / day ;
* Immunosuppression: Any immunosuppressive drugs must be stopped ≥ 4 weeks before enrollment; 9. Volunteer to participate in the clinical trial and sign the informed consent.

Exclusion Criteria:

1. Pregnant or breastfeeding women;
2. Hepatitis B surface antigen (HBsAg) positive; Hepatitis B core antibody (HBcAb) positive, and HBV DNA copy number positive; Hepatitis C antibody (HCV-Ab) positive; Anti-Treponema pallidum antibody (TP-Ab) positive; Human immunodeficiency virus antibody (HIV-Ab) positive; Those who meet any of the following conditions;
3. Any active infection requiring antibiotic treatment;
4. Received any immune cell therapy within one year;
5. Previously received Claudin18.2 targeted therapy ;
6. Live vaccine or live attenuated vaccine received within 4 weeks before single collection;
7. Surgery has been performed within 2 weeks before apheresis and the researchers believe that it may affect the patient's safety;
8. Active coronary heart disease (including angina pectoris, myocardial infarction) within 6 months before enrollment;
9. Within 6 months before study entry, the subject had a history of clinically significant arrhythmias or current abnormalities requiring antiarrhythmic treatment other than beta-blockers or digoxin and/or conduction drugs, excluding atrial fibrillation and paroxysmal supraventricular tachycardia;
10. Left ventricular ejection fraction (LVEF) <50% or congestive heart failure (New York Heart Association NYHA classification ≥3) at screening;
11. Uncontrolled diabetes (glycosylated hemoglobin>8%), uncontrolled hypertension (systolic blood pressure/diastolic blood pressure>160mmHg/100mmHg while taking medication);
12. Patients with active autoimmune diseases within 3 months before screening, such as systemic lupus erythematosus, who need to continue taking medication during the entire trial period;
13. Other malignancies occurred within 5 years before enrollment, excluding cervical carcinoma in situ, skin squamous cell carcinoma, or basal cell carcinoma that had been treated with radical cure;
14. Have a known symptomatic central nervous system (CNS) disease;
15. Tumor cells infiltrate the central nervous system, and tumor cells are detected in the cerebrospinal fluid or the tumor is detected by cranial imaging;
16. The tumor has extensive metastasis and involves more than two organs at the same time, which the investigator believes may significantly change the baseline assessment; or the tumor has progressed rapidly and has reached PD between enrollment and lymph node clearance;
17. Difficult airway (tumor growth blocking the airway or airway deformity, etc.);
18. before apheresis, lymph node ablation, and XKDCT 225 cell injection to maintain fingertip blood oxygen saturation > 95%;
19. The subject has unstable or active gastric ulcer or active gastrointestinal bleeding, or other conditions that may require emergency treatment during the trial, including but not limited to gastrointestinal obstruction, perforation, and rupture of giant tumors;
20. Patients with pleural and abdominal effusion greater than grade 2 during screening and unable to be controlled by drainage or diuretics;
21. The subject is currently taking anticoagulants and cannot stop taking them during the entire trial;
22. Allergy or intolerance to the research drugs tocilizumab, fludarabine, cyclophosphamide and other lymphoproliferative drugs selected by the investigator;
23. Those who are allergic to common emergency and anesthetic drugs, and have life-threatening allergic reactions, hypersensitivity reactions, or intolerance to XKDCT 225 cell preparations or their components; Patients who were deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 28 days of single infusion
  Dose limiting toxicity (DLT) in the dose escalation phase
Maximum tolerated dose (MTD) | 28 days of single infusion
  Maximum tolerated dose (MTD) in the dose escalation phase
The incidence and severity of adverse events (AEs) (%) | 1 year
  The incidence and severity of AEs

SECONDARY OUTCOMES:
Pharmacokinetics (the number of CAR copies (copies/μg gDNA) in peripheral blood) | 1 year
  The number of CAR copies (copies/μg gDNA) were detected by qPCR method to determine the peak time (day) of XKDCT225, sustained survival period (day).
Peripheral blood cytokines | 1 year
  Including IL-6 concentration (pg/ml) , etc.
XKDCT293 immunogenicity assay | 1 year
  employing a validated electrochemiluminescence (ECL) assay on the MESO QuickPlex SQ 120 system from Meso Scale Discovery (MSD). This assay detects XKDCT293 antibody titer (ng/ml) by measuring the emitted light from the SULFO-TAG label.
Objective response rate (ORR) (%) | 1 year
  According to RECIST 1.1 criteria, the percentage of the analyzed population with the best efficacy evaluation reaching CR and PR.
Time to response (TTR) (month) | 1 year
  According to RECIST 1.1 criteria, the time interval from the date of initial infusion of the study drug to the date of initial assessment of partial remission or better outcome in patients with the best efficacy evaluation as partial remission or better outcome.
Duration of Overall Response (DOR) (month) | 1 year
  According to RECIST 1.1 criteria, in patients with the best efficacy evaluation of CR or PR, the time (month) from the first evaluation of the tumor as CR or PR to the first evaluation as PD or death from any cause (whichever occurs first).
Progression-free survival (PFS) (month) | 1 year
  From the first infusion of the study drug to the date of the first recorded tumor progression (whether treated or not) or the date of death for any reason, whichever occurs first.
Overall survival (OS) (month) | 1 year
  The time between the patient's first infusion of the study drug and the patient's death due to various reasons.

CONTACTS AND LOCATIONS:
Locations (1):
- AnYang Tumor Hospital, Anyang, Henan, China

IPD SHARING:
Plan to Share IPD: No